CLINICAL TRIAL: NCT00082836
Title: A Pilot Study of Radiolabeled Indium-111 and Yttrium-90 Ibritumomab Tiuxetan in Primary CNS Lymphoma
Brief Title: Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Recurrent Primary CNS Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 04-009; MSKCC-04009
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab and yttrium Y 90 ibritumomab tiuxetan, can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells.

PURPOSE: This clinical trial is studying how well giving yttrium Y 90 ibritumomab tiuxetan together with rituximab works in treating patients with recurrent primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the absorbed radiation doses of CNS lesions after administration of indium In 111 ibritumomab tiuxetan (for imaging) in patients with recurrent primary CNS lymphoma.

Secondary

* Determine the safety of a therapeutic dose of yttrium Y 90 ibritumomab tiuxetan in these patients.

Tertiary

* Determine the radiographic response in patients treated with this drug.

OUTLINE: Patients receive rituximab IV on day 1. Within 4 hours after rituximab administration, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes. Patients then undergo whole body imaging. Patients whose dosimetry indicates that their CNS lesion would receive a sufficient radioimmunotherapy dose receive a therapeutic dose of yttrium Y 90 ibritumomab tiuxetan IV over 20-30 minutes on day 7.

Patients are followed monthly for 3 months, every 3 months for 2 years, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma (NHL)

  * Recurrent disease

    * Isolated CNS relapse of systemic NHL allowed
  * Primary CNS lymphoma
* Measurable gadolinium-enhancing lesion on MRI of the brain
* No impaired bone marrow reserve
* No hypocellular bone marrow
* No marked reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid)
* No pleural effusion
* No chronic lymphocytic leukemia
* No AIDS-related lymphoma

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Platelet count > 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL

Other

* HIV negative
* No serious nonmalignant disease that would preclude study participation
* No infection
* No anti-murine antibody reactivity*
* No human anti-mouse antibodies
* Not pregnant
* Negative pregnancy test NOTE: *Results must be available prior to study entry for patients who received prior murine antibodies or proteins, other than rituximab

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Radiotherapy
* No prior stem cell transplantation
* No prior myeloablative therapies with autologous bone marrow transplantation or peripheral blood stem cell rescue
* No prior failed stem cell collection
* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* No more than 1 prior chemotherapy regimen

Endocrine therapy

* Not specified

Radiotherapy

* No prior radioimmunotherapy
* No prior whole-brain radiotherapy
* No prior external beam radiotherapy (involved field or regional) to > 25% of active bone marrow

Surgery

* More than 4 weeks since prior major surgery except diagnostic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Dosimetry at 1, 24, and 48 hours

SECONDARY OUTCOMES:
Safety by NCI common toxicty criteria
Radiographic response at 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E. Abrey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States